CLINICAL TRIAL: NCT07143929
Title: An Open-label, Dose-escalation Early-phase Clinical Study of CD7-targeted CAR-T Cells for the Treatment of Relapsed or Refractory Peripheral T Cell Lymphoma (PTCL)
Brief Title: To Observe the CD7-targeted CAR-T Therapy in the Treatment of r/r PTCL
Acronym: S101P
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Anti CD7 CAR-T for r/r PTCL
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: CD7 Positive R/R PTCL

STUDY DESIGN:
Intervention Model Description: 3+3 dose escalation design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti CD7 CAR-T cells (Experimental): eligible patients will be treated with CD7-targeted CAR-T cells
  Interventions: Drug: CAR-T

INTERVENTIONS:
Drug: CAR-T — autologous CD7-targeted CAR-T cells, single injection

SUMMARY:
To observe the efficacy and safety of CD7-targeted chimeric antigen receptor T cells in the treatment of refractory or relapsed PTCL.

DETAILED DESCRIPTION:
In this study, anti CD7 CAR-T cell therapy will be explored for patients with relapsed/refractory PTCL. In this study, the 3+3 dose climbing mode will be used to explore the safety and efficacy of CAR-T cells in r/r PTCL therapy at different doses. The RP2D dose will be determined after the relevant data is summarized。

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old and<80 years old；
2. According to the clinical practice guidelines for T-cell lymphoma of the National Comprehensive Cancer Network (NCCN) (2022. v2), diagnosis of peripheral T-cell lymphoma；
3. Relapse or refractory peripheral T-cell lymphoma, which has not achieved remission or relapsed after receiving ≥ 1 line of systemic treatment in the past；
4. Histologically confirmed as CD7 positive；
5. According to Lugano2014 standard, enhanced CT before enrollment should indicate at least one evaluable tumor lesion, and PET/CT should show metabolic activity.
6. Blood routine neutrophil count ≥ 1.0×109/L during screening; For individuals without bone marrow invasion, platelet count ≥ 75×109/L, Hb≥80g/L; For individuals with bone marrow invasion, platelet count ≥50×109/L, Hb≥60g/L；
7. Creatinine clearance rate>60ml/min (Cockcroft and Gault formula); serum total bilirubin≤1.5 times the upper limit of normal value, and serum ALT and AST ≤ 3 times the upper limit of normal value range;
8. left ventricular Ejection fraction (LVEF) ≥ 50%.
9. Estimated survival time of over 3 months.
10. ECOG: 0-1.
11. Subjects or their Legal guardian voluntarily participate in the trial and sign the informed consent form.

Exclusion Criteria:

1. Primary cutaneous T-cell lymphoma, including mycosis fungoides (MF) and Sezary syndrome (SS); T-lymphoblastic leukemia/lymphoma（T-ALL/LBL）；
2. Primary central nervous system cell lymphoma, or with active central nervous system invasion；
3. If anti-tumor treatment has been received before infusion, and drugs have not been completely eliminated must be excluded;
4. Individuals with a history of allergies to any component in cellular products.
5. Cardiac function:cardiac dysfunction classified as Class III or IV；Myocardial infarction, cardiac angioplasty or stenting, unstable angina pectoris, or other serious heart disease clinically within 12 months of enrollment；The electrocardiogram indicates that the QT interval is significantly prolonged, and the patient has serious heart disease such as serious arrhythmia in the past.
6. Previous history of craniocerebral trauma, Disorders of consciousness, epilepsy, cerebrovascular ischemia, cerebrovascular hemorrhagic disease, etc.
7. Uncontrolled severe active infections.
8. The subject has a history of other primary cancers, except for the following.
9. Subjects with autoimmune diseases requiring treatment or subjects requiring Immunosuppressive drug treatment.
10. Individuals with graft versus host disease (GvHD) and/or requiring immunosuppressive therapy.
11. Live vaccination within 4 weeks prior to screening.
12. The subject has a history of alcoholism, drug abuse, or mental illness.
13. Individuals with EBV DNA copy numbers greater than the upper limit of normal or positive for EBER; CMV copies greater than the upper limit of normal values; HBV or HCV DNA copy number>the upper limit of normal value, and active syphilis or AIDS and other virus infected persons.
14. Subjects who were receiving systemic hormone treatment before screening and who were judged by the investigator to need long-term use of systemic hormone during treatment (except for inhalation or local use).
15. Individuals who have participated in other clinical trials within the first 4 weeks of screening.
16. Pregnant and lactating women and subjects with Fertility who cannot take effective contraceptive measures (both men and women).
17. Any situation that the researcher believes may increase the risk of the subject or interfere with the test results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
safety: Dose-limiting toxicity | at least 28 days after the CAR-T cells infusion
  Observe the incidence rate of DLT events within 28 days after cell infusion

SECONDARY OUTCOMES:
Efficacy of the anti CD7 CAR-T cells to R/R PTCL | at least 1 year after the CAR-T cells infusion
  Remission rate, remission rate includes complete remission(CR)、partial remission(PR)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided